CLINICAL TRIAL: NCT06314243
Title: The Impact of Pumpkin Seed Oil Supplementation on the Clinical Outcome in Hemodialysis Patients
Brief Title: The Impact of Pumpkin Seed Oil Supplementation on Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Merna Nasry, Demonstrator of Clinical Pharmacy Department, Faculty of pharmacy, Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHDIRB2020110301 REC #241
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2024-07

CONDITIONS: Hemodialysis Patients

STUDY DESIGN:
Intervention Model Description: Design: Prospective, randomized, Open label - controlled clinical trial.
  Patients: A total of 56 patients on regular hemodialysis (HD) will be enrolled in the study. These patients will be randomly allocated into two equal groups:
  * Group 1 (PSO group): consists of 28 patients who will receive one capsule containing 1010 mg PSO once daily for 12 weeks, " Ronkin®, KMT PHARMA, Egypt. "
  * Group 2 (Control group): consists of 28 patients who will not receive the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pumpkin Seed Oil group (Experimental): Group 1 (Pumpkin Seed Oil group): consists of 28 patients who will receive one capsule containing 1010 mg PSO once daily for 12 weeks, " Ronkin®, KMT PHARMA, Egypt. "
  Interventions: Dietary Supplement: Pumpkin Seed Oil " Ronkin®, KMT PHARMA, Egypt. "
- Control group (No Intervention): Group 2 (Control group): consists of 28 patients who will not receive the intervention.

INTERVENTIONS:
Dietary Supplement: Pumpkin Seed Oil " Ronkin®, KMT PHARMA, Egypt. " — Ronkin soft gelatin capsules, each containing 1010 mg of pumpkin seed oil (Latin name: Curcurbita pepo), standardized to contain palmitic acid (8-15%), stearic acid (3-8%), oleic acid (15-35%), linoleic acid (40-65%), and other fatty acids (≤ 2.4%)
  Other Names: Pepon
  Arms: Pumpkin Seed Oil group

SUMMARY:
The goal of this clinical trial is to investigate the effects of Pumpkin Seed Oil (PSO) supplementation on systemic inflammation, oxidative stress, and lipid profile in hemodialysis patients.

The main question it aims to answer is:

• Does PSO have a promising effect on systemic inflammation, oxidative stress, and lipid profile in hemodialysis patients?

Patients on regular hemodialysis who take PSO supplementation will be compared to those who don't to see if PSO supplementation improves their systemic inflammation, oxidative stress, and lipid profile.

DETAILED DESCRIPTION:
This study aims to investigate the effects of PSO supplementation on systemic inflammation, oxidative stress, and lipid profile in hemodialysis patients via assessment of IL-6, MDA, lipid profile, and kidney function tests.

Patients & Methods:

Design: Prospective, randomized, Open label - controlled clinical trial.

Patients: A total of 56 patients on regular hemodialysis (HD) will be enrolled in the study. These patients will be randomly allocated into two equal groups:

* Group 1 (PSO group): consists of 28 patients who will receive one capsule containing 1010 mg PSO once daily for 12 weeks, " Ronkin®, KMT PHARMA, Egypt. "
* Group 2 (Control group): consists of 28 patients who will not receive the intervention.

Setting: Adult Nephrology and Dialysis Unit, Ain Shams University Hospital, Cairo, Egypt.

Blood samples will be taken in the dialysis unit and will be sent to Ain Shams University labs for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients older than 18.
* Patients undergoing regular HD for at least 3 months prior to enrollment.
* Not participate in any other clinical trials.
* Physically stable.

Exclusion Criteria:

* Patients taking antioxidant supplements prior to the study's two-month time frame.
* Patients with autoimmune, liver, cancer diseases and acquired immunodeficiency syndrome (AIDS).
* Sensitivity to pumpkin seed oil.
* Patients taking warfarin.
* History of drug or alcohol abuse.
* Pregnant or breastfeeding women and women with the possibility of getting pregnant.
* Smokers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-09-04 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of PSO supplementation on oxidative stress in hemodialysis patients. | 12 weeks
  To evaluate the effect of PSO supplementation on oxidative stress via measuring malondialdehyde (MDA) as oxidative stress marker.
To evaluate the effect of PSO supplementation on the systemic inflammation in hemodialysis patients. | 12 weeks
  To evaluate the effect of PSO supplementation on the systemic inflammation via measuring interleukin-6 (IL-6) as inflammatory marker.

SECONDARY OUTCOMES:
To evaluate the effect of PSO supplementation on the lipid profile in hemodialysis patients. | 12 weeks
  To evaluate the effect of PSO supplementation on the lipid profile, include triglyceride (TG), total cholesterol (TC), LDL, and HDL measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Adult Nephrology and Dialysis Unit, Ain Shams University Hospital, Cairo, Egypt., Cairo, Egypt